CLINICAL TRIAL: NCT06210399
Title: Effectiveness of Extracorporeal Shockwave Therapy in Patients With Chronic Wounds Hospitalized in a Medium Stay Hospital
Brief Title: Shockwave Therapy in Patients With Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guadarrama Hospital (Other)
Collaborators: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Laura Martín Losada, Nurse Director, Guadarrama Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2023-11-21; First posted 2024-01-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Wound Heal
Keywords: Extracorporeal Shockwave Therapy; Wound healing
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Quasi-Experimental Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Extracorporeal Shockwave Therapy (Experimental): The parameters for shock wave therapy will be: frequency 4-6 Hz, intensity 0.075-0.11 mJ/mm2 (millijoules per millimeter), number of pulses 350+10xcm2 (square centimetre) of wound surface (the number of pulsations is dependent of the surface), with sterile field (sterile gel on the wound and sterile transparent film to cover it). They will be applied by sweeping the surface of the wound and 1 centimetre around it. In each session, the session-specific data notebook and the appearance of side effects (pain, bleeding, others) will be recorded. Subsequently, the conventional healing procedure will be applied, according to the procedures for healing chronic wounds of the Guadarrama Hospital.
  Interventions: Procedure: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Procedure: Extracorporeal Shockwave Therapy — 3 to 6 shock wave treatment sessions will be performed (PiezoWave 2 Control Unit Generator, classification 93/42/EEC class IIb), with a frequency of two sessions per week.

SUMMARY:
Introduction: Chronic wounds are a major health problem with impact in the quality of life of patients, increased their morbidity and mortality, nursing burden, extend the hospital stays, and healthcare costs. Searching how to apply the best care available in wounds, shock wave treatment is found in order to stimulate tissue growth in this type of skin injuries. There are different studies to support this recommendation but also there is variability about of patients, different types of injuries or settings. It is considered that more research studies are needed to maintain this evidence and to explore other settings like the effectiveness in a medium stay hospital.

Objectives: To assess the effectiveness of shockwave treatment to reduce the size of chronic wounds.

Method: A quasi-experimental design will be used. The population under study will include patients admitted in the Functional Recovery Unit who present chronic wounds upon admission. The sample size will be 30 patients. An intentional non-probabilistic sampling will be carried out. Main outcome: decrease the wound size. Sociodemographic variables, personal history, comorbidities, current clinical situation, shock wave treatment variables and its evolution will be collected.

Applicability: In case of findings are better than habitually care, the number of treatments required by the patient would be reduced, the patient's state of health would improve, the risk of infection of the wound decrease, and the comfort and quality of life of patients could improve. The findings may represent a change in clinical practice because they may be used to modify the treatment protocols for chronic wounds at the Guadarrama Hospital and in other similar hospitals. Also, they can contribute to the evidence based care which supports shockwave treatment.

DETAILED DESCRIPTION:
Recruitment: the research team will recruit participants who meet inclusion criteria and do not present exclusion criteria, during the first 48 hours of admission to the functional recovery unit. A member of the team will inform and invite the subject or his or her legal representative to participate in the study. The information sheet will be given to the patient and after accepting, he/she has to sign the specific informed consent for the study and the authorization to take images. At that time, the completion of the Data Collection Notebook will begin, which has been prepared ad hoc by the research team. In order to guarantee the confidentiality of the personal data, they will be coded by dissociating the identifying and personal data from those necessary for the configuration of variables. To this end, the personal identity carry out a coding process of the units of analysis. In the event that the same patient has more than one wound that can be included in the study, a data collection notebook will be used for each wound, indicating its location and using the same coding, because the coding number will be associated with each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older,
* To have a chronic wound classified as:

  * pressure ulcer,
  * ischemic wounds,
  * neuropathic wounds,
  * dehiscence of surgical wounds
  * delayed current of wound healing of more than 6 weeks.
* To sign informed consent.

Exclusion criteria:

* To have signs of infection observed in wound.
* Necrotic tissue.
* Tumor wounds.
* Venous thrombosis.
* Large blood vessels at lesion edges.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Decrease wound size area | All wounds will be measured at the end of the intervention (3 weeks).
  Decrease de size area at the end of the intervention. The surface of the wound will be measured in centimeters (length x width)

SECONDARY OUTCOMES:
To quantify the change in the size of chronic wounds treated with shock waves | at the end of the intervention (3 weeks)
  The surface of the wound will be measured in centimeters. The average of the decrease will be evaluated.
To identify the patients variables related to achieve a lesion reduction equal to or greater than 50% of the surface measured in centimeters (greater success in healing). | at the end of the intervention (3 weeks)
  The demographic (aged, sex) and clinic (urinary incontinence, faecal incontinence, personal history, Barthel Index, Norton Scale, blood albumin, smoking habits, type of wound, location of wound, clinical course) variables will be compared with the main variable
To assess number and types of side effects what patients shows related to the use of low-frequency shockwaves in chronic wounds. | at the end of the intervention (3 weeks)
  Side effects (none, bleeding, skin redness, red spots, vasovagal syncope, paresthesia, hypesthesia, others) will be collected after the sessions.
To assess whether the pain perception due to chronic wounds in patients undergoing the intervention decreases. The pain perception will be measured with Visual Analogue Scale (VAS) or Pain Assesment in Advanced Dementia Scale (PAINAD). | Baseline and during the intervention (up 3 weeks)
  Pain will be assessed baseline and during the shockwave session with Visual Analogue Scale (VAS) or Pain Assesment in Advanced Dementia Scale (PAINAD). The tool will be used depending on the patients' cognitive status. VAS and PAINAD scales measure fron 0 to 10 being 0 without pain and 10 the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Martin, RN, MSc, Principal Investigator — Guadarrama Hospital
Locations (1):
- Laura Martín Losada, Guadarrama, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berta L, Fazzari A, Ficco AM, Enrica PM, Catalano MG, Frairia R. Extracorporeal shock waves enhance normal fibroblast proliferation in vitro and activate mRNA expression for TGF-beta1 and for collagen types I and III. Acta Orthop. 2009 Oct;80(5):612-7. doi: 10.3109/17453670903316793. PMID 19916698
- [Background] Chen YJ, Wang CJ, Yang KD, Kuo YR, Huang HC, Huang YT, Sun YC, Wang FS. Extracorporeal shock waves promote healing of collagenase-induced Achilles tendinitis and increase TGF-beta1 and IGF-I expression. J Orthop Res. 2004 Jul;22(4):854-61. doi: 10.1016/j.orthres.2003.10.013. PMID 15183445
- [Background] Corrales Pérez, JM, Águila Pollo, MC, Vázquez Aguilera, M, Jayne Grantham, S, Ramos Sánchez A, Fernandes Ribeiro AS. (2015) Repercusión de las heridas crónicas en las unidades de rehabilitación funcional. Gerokomos [Internet]. 2015 Sep [citado 2023 Abr 08] ; 26( 3 ): 109-114.
- [Background] Domínguez-Saavedra G, Hernández-Galván JM.(2021) Actualización en el manejo de heridas. Cir Plast. 2021;31(3):124-136. doi:10.35366/103715.
- [Background] Fu M, Sun CK, Lin YC, Wang CJ, Wu CJ, Ko SF, Chua S, Sheu JJ, Chiang CH, Shao PL, Leu S, Yip HK. Extracorporeal shock wave therapy reverses ischemia-related left ventricular dysfunction and remodeling: molecular-cellular and functional assessment. PLoS One. 2011;6(9):e24342. doi: 10.1371/journal.pone.0024342. Epub 2011 Sep 6. PMID 21915315
- [Background] Galiano R, Snyder R, Mayer P, Rogers LC, Alvarez O; Sanuwave Trial Investigators. Focused shockwave therapy in diabetic foot ulcers: secondary endpoints of two multicentre randomised controlled trials. J Wound Care. 2019 Jun 2;28(6):383-395. doi: 10.12968/jowc.2019.28.6.383. PMID 31166864
- [Background] GNEAUPP (2019). Prevention and Treatment of Pressure Ulcers/Injuries: Quick Reference Guide 2019 - GNEAUPP
- [Background] Holsapple JS, Cooper B, Berry SH, Staniszewska A, Dickson BM, Taylor JA, Bachoo P, Wilson HM. Low Intensity Shockwave Treatment Modulates Macrophage Functions Beneficial to Healing Chronic Wounds. Int J Mol Sci. 2021 Jul 22;22(15):7844. doi: 10.3390/ijms22157844. PMID 34360610
- [Background] Keil H, Mueller W, Herold-Mende C, Gebhard MM, Germann G, Engel H, Reichenberger MA. Preoperative shock wave treatment enhances ischemic tissue survival, blood flow and angiogenesis in a rat skin flap model. Int J Surg. 2011;9(4):292-6. doi: 10.1016/j.ijsu.2011.01.003. Epub 2011 Jan 21. PMID 21256991
- [Background] Larking AM, Duport S, Clinton M, Hardy M, Andrews K. Randomized control of extracorporeal shock wave therapy versus placebo for chronic decubitus ulceration. Clin Rehabil. 2010 Mar;24(3):222-9. doi: 10.1177/0269215509346083. Epub 2010 Feb 15. PMID 20156981
- [Background] Mittermayr R, Antonic V, Hartinger J, Kaufmann H, Redl H, Teot L, Stojadinovic A, Schaden W. Extracorporeal shock wave therapy (ESWT) for wound healing: technology, mechanisms, and clinical efficacy. Wound Repair Regen. 2012 Jul-Aug;20(4):456-65. doi: 10.1111/j.1524-475X.2012.00796.x. Epub 2012 May 29. PMID 22642362
- [Background] Mittermayr R, Hartinger J, Antonic V, Meinl A, Pfeifer S, Stojadinovic A, Schaden W, Redl H. Extracorporeal shock wave therapy (ESWT) minimizes ischemic tissue necrosis irrespective of application time and promotes tissue revascularization by stimulating angiogenesis. Ann Surg. 2011 May;253(5):1024-32. doi: 10.1097/SLA.0b013e3182121d6e. PMID 21372687
- [Background] National Pressure Injury Alliance, (2019). Guia_.consulta.rapida.LPP_.Spanish.pdf (gneaupp.info) European Pressure Ulcer Advirory. Panel, National Pressure Injury Alliance. Preveión y tratamiento de las leciones/úlceras por presión. Guía de consulta rápida (edición en español)(2019). Emily Haesler
- [Background] Ottomann C, Hartmann B, Tyler J, Maier H, Thiele R, Schaden W, Stojadinovic A. Prospective randomized trial of accelerated re-epithelization of skin graft donor sites using extracorporeal shock wave therapy. J Am Coll Surg. 2010 Sep;211(3):361-7. doi: 10.1016/j.jamcollsurg.2010.05.012. Epub 2010 Jul 14. PMID 20800193
- [Background] Ottomann C, Stojadinovic A, Lavin PT, Gannon FH, Heggeness MH, Thiele R, Schaden W, Hartmann B. Prospective randomized phase II Trial of accelerated reepithelialization of superficial second-degree burn wounds using extracorporeal shock wave therapy. Ann Surg. 2012 Jan;255(1):23-9. doi: 10.1097/SLA.0b013e318227b3c0. PMID 21775883
- [Background] Oyebode OA, Jere SW, Houreld NN. Current Therapeutic Modalities for the Management of Chronic Diabetic Wounds of the Foot. J Diabetes Res. 2023 Feb 10;2023:1359537. doi: 10.1155/2023/1359537. eCollection 2023. PMID 36818748
- [Background] Ramon S, Espanol A, Yebra M, Morillas JM, Unzurrunzaga R, Freitag K, Gomez S, Aranzabal JR. [Current evidences in shockwave treatment. SETOC (Spanish Society of Shockwave Treatment) recommendations]. Rehabilitacion (Madr). 2021 Oct-Dec;55(4):291-300. doi: 10.1016/j.rh.2021.02.002. Epub 2021 Mar 17. Spanish. PMID 33743978
- [Background] Rassweiler JJ, Scheitlin W, Goezen AS, Rassweiler-Seyfried MC. Low-energy Shockwave Therapy in the Management of Wound Healing Following Fournier's Gangrene. Eur Urol Open Sci. 2022 Sep 13;45:8-11. doi: 10.1016/j.euros.2022.08.019. eCollection 2022 Nov. PMID 36131850
- [Background] RNAO. (2016). Valoración y manejo de las lesiones por presión para equipos interprofesionales (Internet) Disponible en: Pressure_Injuries_Spanish BPG.pdf
- [Background] Schaden, W., Kölpl, C., Valentin, A., Pusch, M., & Thiele, R. (2005). Extracorporeal shockwave therapy for chronic skin lesions. In 8th International Congress of the ISMST, May 29th-June 1st (pp. 62-68).
- [Background] Taheri P, Shahbandari M, Parvaresh M, Vahdatpour B. Extracorporeal Shockwave Therapy for Chronic Venous Ulcers: A Randomized Controlled Trial. Galen Med J. 2021 Apr 25;10:e1931. doi: 10.31661/gmj.v10i0.1931. eCollection 2021. PMID 35434156
- [Background] Wang CJ, Wang FS, Yang KD, Weng LH, Hsu CC, Huang CS, Yang LC. Shock wave therapy induces neovascularization at the tendon-bone junction. A study in rabbits. J Orthop Res. 2003 Nov;21(6):984-9. doi: 10.1016/S0736-0266(03)00104-9. PMID 14554209
- [Background] Zhang L, Weng C, Zhao Z, Fu X. Extracorporeal shock wave therapy for chronic wounds: A systematic review and meta-analysis of randomized controlled trials. Wound Repair Regen. 2017 Aug;25(4):697-706. doi: 10.1111/wrr.12566. Epub 2017 Oct 18. PMID 28759136